CLINICAL TRIAL: NCT05565196
Title: Implementing the Birth Companion Intervention Package in Ethiopia, Kenya and Nigeria: Feasibility, Acceptability, and Impact on Coverage of Facility Births Attended by a Companion.
Brief Title: Birth Companion Intervention in Ethiopia, Kenya and Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Addis Continental Institute of Public Health (Other); St Paul's Hospital Millennium Medical College (Unknown); International Center for Reproductive Health Kenya (Unknown); Bill and Melinda Gates Foundation (Other); Maternal and Reproductive Health Research Collective (Unknown)
Responsible Party: Principal Investigator, Della Berhanu, Research lead, Jhpiego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00021183
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-04

CONDITIONS: Maternal Care Patterns

STUDY DESIGN:
Masking Description: 6801
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Birth companion intervention arm (Experimental): Women who deliver in facilities in the experimental arm will be exposed to a facility-based intervention designed to improve companionship in labor, childbirth, and postpartum periods.
  Interventions: Behavioral: Birth companions
- Standard of care arm (No Intervention): Women who deliver in facilities in the experimental arm will be exposed to the standard of care for labor, delivery, and the postpartum period.

INTERVENTIONS:
Behavioral: Birth companions — The intervention will have the following components: 1) Orient facilities and providers to benefits of BC; 2) Develop/update formal standard operating procedures (SOP) for implementing BC and develop plans to implement SOP; 3) Assess data required for implementation and an audit and feedback cycle for tracking coverage; 4) Assess and carry out modest structural changes in facilities to facilitate BC; 5) Use human centered design to develop materials/resources and a means to distinguish/recognize the BC, taking into account common barriers and misconceptions; 6) Prepare providers to integrate BC into care team; 7) Orient ANC clients to BC rationale and selection; 8) Prepare BCs to support women; 9) Iterate model and track intervention/policies.
  Arms: Birth companion intervention arm

SUMMARY:
The study aims to assess the acceptability; feasibility; implementation cost; and penetration of the birth companion intervention introduced at health facilities. It is a multi-country study (Ethiopia, Kenya and Nigeria) with a two parallel arm cluster randomized controlled trial design. The study duration will approximately be 16 months.

DETAILED DESCRIPTION:
The overall purpose of this study is to investigate how a birth companion (BC) intervention can be implemented to increase the proportion of women who are accompanied by a BC during labor, childbirth, and postpartum in Ethiopia, Kenya and Nigeria. After baseline data collection, facilities will be randomized in a 3:1 ratio; for every three facilities that receive the BC intervention, one facility will serve as a control facility. After randomization, over the course of two months, intervention facilities will start preparing to introduce the BC intervention to facilitate presence of BC during labor and delivery, while the control facilities will continue to provide the local standard of routine care. The intervention will have the following components: 1) Orient facilities and providers to benefits of BC; 2) Develop/update formal standard operating procedures (SOP) for implementing BC and develop plans to implement SOP; 3) Assess data required for implementation and an audit and feedback cycle for tracking coverage; 4) Assess and carry out modest structural changes in facilities to facilitate BC; 5) Use human centered design to develop materials/resources and a means to distinguish/recognize the BC, taking into account common barriers and misconceptions; 6) Prepare providers to integrate BC into care team; 7) Orient antenatal care (ANC) clients to BC rationale and selection; 8) Prepare BCs to support women; 9) Iterate model and track intervention/policies. Investigators will use a mixed methods approach to address the implementation research questions with exit interviews, health facility register data extraction, in-depth interviews, focus group discussions, and key informant interviews. Investigators will collect quarterly quantitative and qualitative data over the course of one week each, for a total of five data collection periods including baseline.

ELIGIBILITY:
Inclusion Criteria:

Facilities

* Prior to randomization, head of facility grants permission for facility to participate in the study
* Be willing to develop, adopt, and implement the BC standard operating procedures and other components of the BC intervention package
* Have more than 16 births per month during the past three months
* Be in the Addis Ababa and surrounding area, Ethiopia, in Muranga and Machakos County, Kenya or Nasarawa and Kano states, Nigeria

Providers

* At the time of enrollment, providers need to work in ANC or labor and delivery ward(s) of the study facilities
* Able and willing to provide informed consent to participate in the study

Mothers

* Per participant report, age 15 years or older
* Have vaginal birth
* Able and willing to provide informed consent to participate in the study

Birth companions

* Per participant report, for emancipated minors, age 15 years or older. If not an emancipated minor, per participant report, 18 years or older
* Was present at labor and/or delivery
* Identified as a BC by the delivering mother
* Able and willing to provide informed consent to participate in the study

Unit managers

* Involved in the implementation and management of the BC intervention
* Able and willing to provide informed consent to participate in the study

Exclusion Criteria:

Facilities

* Facility staff strike or other disturbance to routine care noted prior to randomization that would pose significant challenge(s) to achieving the study objectives

Providers

* N/A

Mothers

* Unable to participate in an interview due to their physical or emotional condition caused by an adverse delivery outcome.
* Unable to provide valid information because of mental or other serious health condition

Birth companions

* Unable to provide valid information because of mental or other serious health condition

Unit managers

* N/A

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10360 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change in Birth Companion Coverage | Between baseline and Endline survey (12 months after intervention is initiated).
  Between baseline and endline surveys, the investigators will measure the change in the proportion of women who are accompanied by a birth companion during labor, childbirth, and postpartum.

SECONDARY OUTCOMES:
Choice of Birth Companion | Between baseline and Endline survey (12 months after intervention is initiated).
  Between baseline and endline surveys, among women who report having a birth companion, the investigators will measure the change in the proportion who report that their birth companion was the one of their choice.
Change in Experience of Care (Mothers'-Quantitative) | Between baseline and Endline survey (12 months after intervention is initiated).
  Between baseline and endline surveys, the investigators will measure the change in mothers' score on Person-Centered Maternity Care scale. This scale has 33 items with a score ranging from 0-98. A low score signifies a better outcome.
Experience of Care (Mothers'-Qualitative) | Quarterly after initiation of the intervention (for a period of 12 months).
  In intervention facilities, among women who had birth companions investigators will use in-depth interviews to explore their perception of having a birth companion.
Feasibility (Unit managers and Providers-Quantitative) | Endline survey (12 months after intervention is initiated).
  In intervention facilities, investigators will measure the proportion of providers and unit managers who report the physical environment of care supports the presence of birth companions during labor, birth, and the postnatal period.
Feasibility (Unit Managers-Qualitative) | Quarterly after the initiation of the intervention (for a period of 12 months).
  In intervention facilities, investigators will use key informant interviews to understand unit managers' perception on the feasibility of having birth companions.
Acceptability (Mothers) | Quarterly after the initiation of the intervention (for a period of 12 months).
  In intervention facilities, investigators will use in-depth interviews to understand mothers' perception on the acceptability of having birth companions.
Acceptability (Birth Companions) | Quarterly after the initiation of the intervention (for a period of 12 months).
  In intervention facilities, investigators will use in-depth interviews to understand birth companions' perception on the acceptability of being a birth companion.
Acceptability (Providers) | Quarterly after the initiation of the intervention (for a period of 12 months).
  In intervention facilities, investigators will use focus group discussions to understand providers' perception on the acceptability of having birth companions.
Acceptability (Unit Managers) | Quarterly after the initiation of the intervention (for a period of 12 months).
  In intervention facilities, investigators will use qualitative methods understand unit managers' perception on the acceptability of having birth companions.

OTHER OUTCOMES:
Potential association between baseline facility readiness and intervention coverage | Endline survey (12 months after intervention is initiated)
  In intervention facilities, investigators will measure score on facility readiness to change (at baseline) to explore potential association with coverage of the intervention at endline. The tool used for facility staff has scale with 19 items and the score ranges from 0 to 57. The tool used for facility leaders has a scale with 34 items and a score ranging from 0 to 100. Low score means better outcome.
Cost | Endline survey (12 months after intervention is initiated)
  In intervention facilities investigators will collect data on facility-level costs for updates to physical environment of care and other implementation costs.

CONTACTS AND LOCATIONS:
Locations (5):
- Saint Paul's Millennium College, Addis Ababa, Ethiopia
- Kenya (2):
  - Machakos County Health Office, Machakos
  - Murang'a County Health Office, Murang’a
- Nigeria (2):
  - Kano State Health Office, Kano
  - Nasarawa Sate Health Office, Karu

IPD SHARING:
Plan to Share IPD: No
Per current Bill & Melinda Gates Foundation policy for study data

REFERENCES:
- [Derived] Berhanu D, Bekele G, Melesse H, Taddese F, Owira P, Manguro G, Laleye O, Farouk Z, Balogun M, Hyre A, Mwaura S, Kiptoo OK, Wabwile VM, Mohammed S, Wolde K, Teno D, Eke EC, Don-Aki JO, Noguchi L, Suhowatsky S, Doggett E, Yenokyan G, Worku A. A clustered randomized control trial to assess feasibility, acceptability, and impact of implementing the birth companion intervention package in Ethiopia, Kenya, and Nigeria: study protocol. BMC Health Serv Res. 2023 Oct 14;23(1):1100. doi: 10.1186/s12913-023-10082-w. PMID 37838662